CLINICAL TRIAL: NCT04499456
Title: Analysis of Mediators and Moderators of a Web-based Intervention for Alcohol Use Among College Students
Brief Title: Mediators and Moderators of a Web-based Intervention for Alcohol Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, André Bedendo, Sponsor-Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/13831-9
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Waiting list control receiving the PNF after the last assessment
  Interventions: Other: Personalised Normative Feedback
- Single PNF (Experimental): Receives PNF after the first assessment only
  Interventions: Other: Personalised Normative Feedback
- Boosted PNF (Experimental): Receives PNF after every assessment
  Interventions: Other: Personalised Normative Feedback

INTERVENTIONS:
Other: Personalised Normative Feedback — The Personalised Normative Feedback provides information on 1) alcohol consumption (the number of drinks consumed, alcohol-pattern use, binge drinking); 2) normative comparisons; 3) alcohol-related consequences; 4) practical costs of alcohol consumption (money spent and calories consumed); 5) strategies to avoid or risks associated with alcohol use.

SUMMARY:
Background: Alcohol use among college students causes health and social problems. However, even when available, many students do not access alcohol interventions. Web-based Personalized Normative Feedback (PNF) has been used to disseminate alcohol brief-interventions, and evidence supports PNF efficacy in reducing alcohol consumption among this population. On the other hand, studies on PNF mediators and moderators are scarce, limiting the knowledge on the mechanisms of change and conditions in which their effects occur. Objective: to evaluate whether normative perceptions mediate, and motivation to receive the intervention, moderates the effects of a web-based PNF intervention (Pesquisa Universitária sobre Bebidas - PUB 2.0) for alcohol use among Brazilian college students. Methods: Pragmatic randomized controlled trial among college students aged 18 and over and with follow-up assessments after 1, 3 and 6 months. Participants will be randomized into a Control group (assessment only) or to receive the updated version of the intervention (PUB 2.0). Outcomes are the typical number of drinks (primary outcome) and the total number of drinks consumed, drinking frequency, maximum number of drinks consumed and number of consequences (secondary outcomes). Statistical analyses will consider Structural Equation Models and significance level of 5%. This study will improve knowledge on how and in which conditions a web-based alcohol PNF effects occur, helping tailor future strategies to reduce the impact of alcohol problems among college students.

ELIGIBILITY:
Inclusion Criteria:

* College student
* Alcohol use during the last year
* Aged 18 or more years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 685 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Typical alcohol use | 30 days
  The number of typical drink units consumed
Maximum alcohol use | 30 days
  The number of maximum drink units consumed

SECONDARY OUTCOMES:
Frequency of alcohol use | 30 days
Total number of drink units | 30 days
Number of consequences | 30 days
  The number of consequences

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Psicobiologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided